CLINICAL TRIAL: NCT00878696
Title: Influence of Tonic and Burst TMS Characteristics on Acute Inhibition of Subjective Tinnitus
Brief Title: Influence of Tonic and Burst Transcranial Magnetic Stimulation (TMS) Characteristics on Acute Inhibition of Subjective Tinnitus
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof Van de Heyning, UZA
Other Study IDs: ITBTMS
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tinnitus: Tinnitus patients
  Interventions: Procedure: TMS transcranial magnetic stimulation

INTERVENTIONS:
Procedure: TMS transcranial magnetic stimulation — 200 pulses of tonic TMS (see Graph 1) were administered with an intensity at 50% of the maximal TMS device output (50%DO).
  The frequency of the tonic pulses was randomly chosen between 1Hz, 5Hz, 10Hz or 20Hz.
  Burst stimulation was delivered at a burst frequency of 5, 10 or 20Hz. Each burst consisted of 3, 5 or 10 pulses. The individual pulse rate within a burst was 50 or 100Hz.

SUMMARY:
Transcranial magnetic stimulation (TMS) is already broadly used in different areas of neuroscience research. Last year, special attention was drawn to TMS in tinnitus. The aim of the researchers' study is to investigate the stimulation characteristics of TMS in tinnitus patients, in particularly the effect of tonic and burst stimulation of the superior temporal lobe.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to our Multidisciplinary Tinnitus Clinic with tinnitus as a main complaint.

Exclusion Criteria:

* Patients with known history of epilepsy, pacemakers, cochlear implants, neurostimulators or intracerebral pathology were excluded from the study.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented to our Multidisciplinary Tinnitus Clinic with tinnitus as a main complaint.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
VAS visual analogue scale | immediately before and immediately after single session TMS

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium